CLINICAL TRIAL: NCT04069533
Title: A Phase II Clinical Trial to Evaluate the Efficacy of the Infusion of Autologous CD34+ Cells Transduced With a Lentiviral Vector Carrying the FANCA Gene (Orphan Drug) in Patients With Fanconi Anemia Subtype A
Brief Title: Lentiviral-mediated Gene Therapy for Pediatric Patients With Fanconi Anemia Subtype A
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP-L102-0118; 2018-002502-31 (EudraCT Number)
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Fanconi Anemia Complementation Group A
Keywords: anemia; bone marrow failure; gene therapy
MeSH Terms: conditions — Fanconi Syndrome; Anemia; Bone Marrow Failure Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- RP-L102 (Experimental): RP-L102 is CD34+ enriched cells from subjects with Fanconi anemia subtype A transduced ex vivo with lentiviral vector carrying the FANCA gene
  Interventions: Biological: RP-L102

INTERVENTIONS:
Biological: RP-L102 — CD34+ enriched cells from subjects with Fanconi anemia subtype A transduced ex vivo with lentiviral vector carrying the FANCA gene

SUMMARY:
This is an open-label Phase II clinical trial to evaluate the efficacy of a hematopoietic cell-based gene therapy for pediatric patients with Fanconi Anemia, subtype A (FA-A).

Hematopoietic stem cells from mobilized peripheral blood of patients with FA-A will be transduced ex vivo (outside the body) with a lentiviral vector carrying the FANCA gene. After transduction, the corrected stem cells will be infused intravenously back to the patient with the goal of preventing bone marrow failure.

DETAILED DESCRIPTION:
This is a pediatric open-label Phase II clinical trial to assess the efficacy of a hematopoietic gene therapy consisting of autologous CD34+ enriched cells transduced with a lentiviral vector carrying the FANCA gene in pediatric subjects with FA-A.

Enriched CD34+ hematopoietic stem cells will be transduced ex vivo with the therapeutic lentiviral vector and infused via intravenous infusion following transduction without any prior conditioning.

ELIGIBILITY:
Inclusion Criteria:

1. Fanconi anemia as diagnosed by chromosomal fragility assay of cultured lymphocytes in the presence of diepoxybutane (DEB) or similar DNA-crosslinking agent
2. Patient of the complementation group FA-A
3. Minimum age: 1 year and minimum weight of 8 kg.
4. Maximum age: 17 years
5. At least 30 CD34+ cells/µL are determined in one BM aspiration within 3 months prior to the CD34+ cell collection.
6. Provide informed consent in accordance with current legislation
7. Women of childbearing age must have a negative urine pregnancy test at the baseline visit, and accept the use of an effective contraception method during participation in the trial

Exclusion Criteria:

1. Patients with an available and medically eligible human leukocyte antigen (HLA)-identical sibling donor
2. Evidence of myelodysplastic syndrome or leukemia, or cytogenetic abnormalities other than those predictive of these conditions in bone marrow (BM) aspirate analysis. This assessment should be made by valid studies conducted within the 3 months before the patient enters the clinical trial
3. Patients with somatic mosaicism associated with stable or improved counts in all PB cell lineages (If T-lymphocyte chromosomal fragility analysis indicates potential mosaicism, a medically significant decrease in at least one blood lineage over time must be documented to enable eligibility)
4. Lansky performance index ≤ 60%
5. Any concomitant disease or condition that, in the opinion of the Principal Investigator, deems the patient unfit to participate in the trial
6. Pre-existing sensory or motor impairment >/= grade 2 according to the criteria of the National Cancer Institute (NCI)
7. Pregnant or breastfeeding women
8. Hepatic dysfunction as defined by either:

   * Bilirubin > 3 x the upper limit of normal (ULN)
   * Alanine aminotransferase (ALT ) > 5 x ULN
   * Aspartate aminotransferase (AST) > 5 x ULN For subjects with bilirubin, ALT, or AST above ULN, a workup to identify the etiology of liver abnormality should be conducted prior to confirmation of eligibility as stipulated in exclusion criterion 5, including evaluation of viral hepatitis, iron overload, drug injury or other causes.
9. Renal dysfunction requiring either hemodialysis or peritoneal dialysis
10. Pulmonary dysfunction as defined by either:

    * Need for supplemental oxygen during the prior 2 weeks (in absence of acute infection)
    * Oxygen saturation (by pulse oximetry) <90%
11. Evidence of active metastatic or locoregionally advanced malignancy for which survival is anticipated to be less than 3 years
12. Subject is receiving androgens (i.e. danazol, oxymetholone)
13. Subject is receiving other investigational therapy for treatment/prevention of FA-associated bone marrow failure

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Phenotypic correction of bone marrow colony forming units after infusion of RP-L102 | 3 years
  During months 12-36 post-infusion, the survival of bone marrow colony forming units to 10nM mitomycin C (MMC) increases to over or equal to 10% with respect to values determined at baseline (pretreatment evaluation).

SECONDARY OUTCOMES:
Phenotypic correction of T-lymphocytes in peripheral blood after infusion of RP-L102 | 3 years
  Assessment of the percentage of peripheral blood T-cells with diepoxybutane (DEB)-induced chromosomal aberrations that decreases from over or equal to 50% at baseline (defined as the interval between the pre-treatment evaluation and 2 months post-infusion) to less than 50% during the interval between 12 and 36 months post-infusion.
Engraftment of gene-corrected hematopoietic cells after infusion of RP-L102 | 3 years
  The level of gene marking of the FANCA-lentiviral vector (LV) provirus in total peripheral blood cells is at least 0.1 vector copy number (VCN) in peripheral blood cells during months 6-36 post-infusion.
Prevention or rescue of bone marrow failure | 3 years
  Assessment of the need for treatment of bone marrow failure.
Short- and long-term Safety | 3 years
  Evaluation of the number of RP-L102 related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Julián Sevilla Navarro, MD, PhD, Principal Investigator — Hospital Infantil Universitario Niño Jesús (HIUNJ)
Locations (2):
- Hospital Infantil Universitario Niño Jesús (HIUNJ), Madrid, Spain
- University College London Great Ormond Street Institute of Child Health (GOSH), London, United Kingdom